CLINICAL TRIAL: NCT04851210
Title: Identification of miRNAs Associated With Gender Difference in Osteoarthritis Patients
Acronym: MIRGOA
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 148/2021/Sper/IOR
Record Dates: First submitted 2021-04-13; First posted 2021-04-20 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis
Keywords: miRNA; osteoarthritis; gender; biomarker
MeSH Terms: conditions — Osteoarthritis; Coitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and synovial fluid specimen, surgical waste joint tissues (bone, sinovia, cartilage)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The biological study involves the collection of samples from male and female patients (intraoperative waste tissue, blood and synovial fluid), suffering from mild and moderate-severe OA, who undergo endo or arthro-prosthesis surgery, or arthroplasty, for the identification and characterization of a panel of "gender-specific" miRNAs. MicroRNAs will be extracted from the samples (chondrocytes, synoviocytes, osteoblasts and plasma) and will be molecularly characterized in order to identify a panel of miRNAs differently expressed according to the gender and severity of OA. The lymphocyte and phenotypically and functionally characterized populations will be isolated from the corpuscular component and the synovial fluid, in order to evaluate a possible gender-specific difference in the progression of OA-dependent inflammation.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a chronic degenerative joint disease of considerable socio-economic impact, of which a primary and a secondary form are distinguished. Primary OA is a mild form that occurs mainly in the joints of the hands, feet, knee, and hip, and appears in young subjects. Secondary OA derives from different factors that modify the microenvironment of the cartilage such as trauma, congenital joint deformities, metabolic defects, infections that cause post-infectious arthritis, endocrine and neuropathic diseases and disorders that alter the normal structure and function of hyaline cartilage (eg . rheumatoid arthritis, gout, chondrocalcinosis), and is more prevalent in old age.

As regards the secondary form of OA, correlated with advancing age due to the natural aging process of the joint and to events of a traumatic nature, it is hypothesized that a key role in the etiology and progression of the disease may be played by the genre. Immune responses are known to differ in males and females. Some meta-analyzes reveal how the presence of some polymorphisms (ADAM12) in male patients predispose to the development of OA more than in women, especially in the knee joint. Furthermore, new molecular evidence suggests that in patients with OA there is a gender-specific activation of PI3K-AKT and hypoxia signaling, suggesting the presence of possible gender-specific protein factors that may modulate bone metabolism and disease progression. In this regard, studies evaluating the responses of joint chondrocytes to systemic factors suggest that there are differences in the biochemical and molecular characteristics of male and female cells, without prejudice to the fundamental role of hormones in the different gender-specific response to the development and progression of pathology.

It is widely known that the regulation of bone remodeling processes is entrusted to a hormonal mechanism, which mainly involves parathyroid hormone, vitamin D and calcitonin. Other hormone regulators involved are sex hormones (estrogen, testosterone), thyroid hormones, corticosteroids (including cortisone), insulin, and growth factors (including growth hormone).

In the development of OA it is thought that sex hormones may act in a prevalent way. In women of childbearing age, estrogen has a protective action on the bone, inhibiting bone remodeling, especially bone resorption; while in the post-menopausal period, circulating estrogens are reduced compared to testosterone, strongly contributing to an imbalance in bone remodeling, favoring the stiffening of the subchondral bone and the development of osteophytes at the joint margins. The osteophytes seem to be developed in an attempt to stabilize the joint damage. Consequently, the synovial membrane becomes inflamed and thickened, producing synovial fluid with less viscosity and in greater quantities and favoring the development of an inflammatory process on site. Obviously, the entire joint will be damaged up to the reduction of joint mobility and ankylosis.

Similarly men, even if they do not undergo a real andropause, starting from 45 years of age they suffer a progressive decline in the production and release of testosterone, whose levels after the age of 65 are no longer sufficient to maintain good efficiency of the bone tissue favoring its resorption and the possible onset of the pathology. However, it is not known whether the potential differences related to gender, in terms of hormonal release and alteration of bone homeostasis, may be related to the severity of the disease, that is to the development of the inflammatory condition associated with it.

It is therefore necessary to highlight another characteristic of OA, both in terms of development and progression, namely the different inflammatory response based on the patient's gender. In OA, as with other inflammatory diseases, the response of the male immune system induced by inflammation of the synovium and synovial fluid is different than in the female counterpart, suggesting that there could be differences between the two sexes in the levels of immunomodulators in joint tissues, including the synovial membrane, synovial fluid and cartilage itself. Recent studies attribute to the inflammatory microenvironment a key role in the prognosis of the disease.

Recently, the investigators obtained evidences regarding the role of microRNAs and lncRNAs as biomarkers of bone regeneration, directly involving specific cellular signalings (hypoxia, epithelium-mesenchyma transition and mechano-transduction), and representing, in some cases, a crucial point for the development of orthopedic diseases, such as osteoporosis, OA and forms of degeneration of the intervertebral discs. From an ongoing screening on tissue (joint) miRNA and lncRNA differently expressed and which could play a key role in the process of osseointegration of the prosthetic implant, miR-31-5p, miR-33a-5p, miR-133a, miR-675-5p and lncH19 were also evaluated. The correlation analysis between their expression profile and the patient's gender show a different expression of some of them and a gender-specific response on target genes and signaling.

The hypothesis of the study is that there are gender differences that contribute to the increase in the incidence and severity of OA, both in molecular terms (qualitative and quantitative differences in miRNAs involved in transcriptional and translational gene regulation) and inflammatory, such as differences in the development and progression of the lymphocyte population, involved in the OA-related inflammatory response. Therefore, the study aims to identify, characterize and evaluate an expression panel of tissue and circulating miRNAs isolated from patients with both mild and moderate-severe OA, who undergo prosthetic surgery, so as to be able to define possible gender-specific biomarkers of disease progression useful for controlling the osteointegration process of the prosthetic implant, and to be correlated with the pre- and post-operative inflammatory response.

The biological study involves the collection of samples from patients of both sexes suffering from OA, be it mild or moderate-severe, who undergo endo or arthro-prosthesis surgery, or arthroscopy. In particular, the following samples will be collected: 1) cells, such as synoviocytes, osteoblasts and chondrocytes deriving from operating waste tissues; 2) synovial fluid isolated during the operation; and 3) peripheral blood, from which to isolate the plasma and the lymphocyte component, taken 24 hours before surgery, and 72 hours and 1 month after surgery.

The miRNAs will be isolated from the samples isolated from tissues and plasma and will be molecularly characterized in order to identify a panel (also built starting from information obtained from the literature) expressed on the basis of the gender and severity of OA. The identified miRNAs will be validated, in vitro, using a specific molecular approach. The lymphocyte component of the blood and, isolated by means of special separation protocols through cell-specific magnetic beads, will be phenotypically characterized by a flow cytometric approach. The lymphocyte populations that will show a different phenotype between the male and female gender in correlation with the aggressiveness of the disease, will be analyzed and monitored over time up to 1 month of follow-up together with the analysis of synovial fluids, through in vitro studies of cytokine release and ELISA assays.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes suffering from OA in hospital for the surgical treatment of OA (endo- or arthroplasty, or arthroscopy) with an interval of at least three months from any previous infiltrative treatment of any kind;
* Patients with a Kellgren and Lawrence (KL) [Kohn 2016] score greater than or equal to grade III will be enrolled in the 'Moderate-severe OA' group and those with grade I and II KL scores in the 'MIld OA' group;
* Patients able to provide the list of medications and supplements taken;
* Patients able to provide informed consent to treatment.

Exclusion Criteria:

* Patients who have undergone previous joint surgery or who have excessive joint deformity.
* Patients with recent trauma, osteonecrosis or OA induced by previous or current joint infection;
* Patients with metabolic pathologies;
* Patients with previous or current oncological pathologies;
* Women in a climacteric (date of last menstruation less than one year);
* Patients with severe cognitive deficits or psychiatric disorders;
* Autoimmune diseases (eg rheumatoid arthritis).

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A maximum number of n = 20 patients with clinical and radiological diagnosis of OA will be enrolled: n = 10 with OA defined as "moderate-severe" equivalent to the KL score greater than or equal to grade III (n = 5 males and n = 5 females); and n = 10 with OA defined as "mild" equivalent to the grade I and II KL score (n = 5 males and n = 5 females), who undergo endo or arthro-prosthesis surgery, or arthroscopy. All patients will be enrolled in the clinical trial only after having personally dated and signed the written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change assessment of OA 'gender-specific miRNA panel during time | Time points: 24 hours; 72 hours; 1 month
  Identification and characterization of a 'gender-specific' miRNA panel related to disease progression in patients with mild OA (OA with Kellgren Lawrence-KL grade I and II) and moderate-severe (OA with greater or greater KL score equal to grade III).
  The miRNAs will be isolated from patients affected by OA who undergo endo- or arthro-prosthesis operations starting: 1) from cells isolated from waste tissues; and 2) from the plasma taken 24 hours before surgery, and subsequently at 72 hours and 1 month from this.

SECONDARY OUTCOMES:
Functional role of OA 'gender-specific' miRNAs | 2 months
  Define the functional role (regulated or modulated signaling) of each deregulated (up or down-regulated) miRNA through specific in vitro studies.
Change assessment of OA 'gender-specific' inflammatory response during time | Time points: 24 hours; 72 hours; 1 month
  Characterize any differences in the inflammatory response (release of cytokines and inflammatory factors) based on the patient's gender and the severity of the disease, analyzing the lymphocyte component isolated from the blood sample performed 24h before and 72h and 1 month after surgery and analyzing the liquid synovial isolated in the operative site.
OA 'gender-specific' miRNAs as biomarkers of osteointegration | 12 months
  Define some miRNAs (modulated in the same way at the tissue and circulating level) that can be used as "gender-specific" predictive biomarkers of the efficiency of the osteointegrative capacity in the patient with OA.

CONTACTS AND LOCATIONS:
Overall Officials: Viviana Costa, B.Sc Ph.D, Principal Investigator — IRCCS Istituto Ortopedico Rizzoli
Locations (1):
- Dipartimento Rizzoli Sicilia - Istituto Ortopedico Rizzoli, Bagheria, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amodio N, Stamato MA, Gulla AM, Morelli E, Romeo E, Raimondi L, Pitari MR, Ferrandino I, Misso G, Caraglia M, Perrotta I, Neri A, Fulciniti M, Rolfo C, Anderson KC, Munshi NC, Tagliaferri P, Tassone P. Therapeutic Targeting of miR-29b/HDAC4 Epigenetic Loop in Multiple Myeloma. Mol Cancer Ther. 2016 Jun;15(6):1364-75. doi: 10.1158/1535-7163.MCT-15-0985. Epub 2016 May 18. PMID 27196750
- [Background] Bellavia D, De Luca A, Carina V, Costa V, Raimondi L, Salamanna F, Alessandro R, Fini M, Giavaresi G. Deregulated miRNAs in bone health: Epigenetic roles in osteoporosis. Bone. 2019 May;122:52-75. doi: 10.1016/j.bone.2019.02.013. Epub 2019 Feb 14. PMID 30772601
- [Background] Costa V, Lo Dico A, Rizzo A, Rajata F, Tripodi M, Alessandro R, Conigliaro A. MiR-675-5p supports hypoxia induced epithelial to mesenchymal transition in colon cancer cells. Oncotarget. 2017 Apr 11;8(15):24292-24302. doi: 10.18632/oncotarget.14464. PMID 28061476
- [Background] Costa V, Raimondi L, Conigliaro A, Salamanna F, Carina V, De Luca A, Bellavia D, Alessandro R, Fini M, Giavaresi G. Hypoxia-inducible factor 1Alpha may regulate the commitment of mesenchymal stromal cells toward angio-osteogenesis by mirna-675-5P. Cytotherapy. 2017 Dec;19(12):1412-1425. doi: 10.1016/j.jcyt.2017.09.007. Epub 2017 Oct 27. PMID 29111380
- [Background] Costa V, Carina V, Conigliaro A, Raimondi L, De Luca A, Bellavia D, Salamanna F, Setti S, Alessandro R, Fini M, Giavaresi G. miR-31-5p Is a LIPUS-Mechanosensitive MicroRNA that Targets HIF-1alpha Signaling and Cytoskeletal Proteins. Int J Mol Sci. 2019 Mar 28;20(7):1569. doi: 10.3390/ijms20071569. PMID 30925808
- [Background] Costa V, Carina V, Raimondi L, De Luca A, Bellavia D, Conigliaro A, Salamanna F, Alessandro R, Fini M, Giavaresi G. MiR-33a Controls hMSCS Osteoblast Commitment Modulating the Yap/Taz Expression Through EGFR Signaling Regulation. Cells. 2019 Nov 22;8(12):1495. doi: 10.3390/cells8121495. PMID 31771093
- [Background] Gago-Fuentes R, Fernandez-Puente P, Megias D, Carpintero-Fernandez P, Mateos J, Acea B, Fonseca E, Blanco FJ, Mayan MD. Proteomic Analysis of Connexin 43 Reveals Novel Interactors Related to Osteoarthritis. Mol Cell Proteomics. 2015 Jul;14(7):1831-45. doi: 10.1074/mcp.M115.050211. Epub 2015 Apr 22. PMID 25903580
- [Background] Hunziker EB. Articular cartilage repair: basic science and clinical progress. A review of the current status and prospects. Osteoarthritis Cartilage. 2002 Jun;10(6):432-63. doi: 10.1053/joca.2002.0801. PMID 12056848
- [Background] Kohn MD, Sassoon AA, Fernando ND. Classifications in Brief: Kellgren-Lawrence Classification of Osteoarthritis. Clin Orthop Relat Res. 2016 Aug;474(8):1886-93. doi: 10.1007/s11999-016-4732-4. Epub 2016 Feb 12. No abstract available. PMID 26872913
- [Background] Kriegova E, Manukyan G, Mikulkova Z, Gabcova G, Kudelka M, Gajdos P, Gallo J. Gender-related differences observed among immune cells in synovial fluid in knee osteoarthritis. Osteoarthritis Cartilage. 2018 Sep;26(9):1247-1256. doi: 10.1016/j.joca.2018.04.016. Epub 2018 May 19. PMID 29753948
- [Background] Lo Dico A, Costa V, Martelli C, Diceglie C, Rajata F, Rizzo A, Mancone C, Tripodi M, Ottobrini L, Alessandro R, Conigliaro A. MiR675-5p Acts on HIF-1alpha to Sustain Hypoxic Responses: A New Therapeutic Strategy for Glioma. Theranostics. 2016 May 8;6(8):1105-18. doi: 10.7150/thno.14700. eCollection 2016. PMID 27279905
- [Background] Lv ZT, Liang S, Huang XJ, Cheng P, Zhu WT, Chen AM. Association between ADAM12 Single-Nucleotide Polymorphisms and Knee Osteoarthritis: A Meta-Analysis. Biomed Res Int. 2017;2017:5398181. doi: 10.1155/2017/5398181. Epub 2017 Aug 8. PMID 28929114
- [Background] Pan Q, O'Connor MI, Coutts RD, Hyzy SL, Olivares-Navarrete R, Schwartz Z, Boyan BD. Characterization of osteoarthritic human knees indicates potential sex differences. Biol Sex Differ. 2016 Jun 2;7:27. doi: 10.1186/s13293-016-0080-z. eCollection 2016. PMID 27257472
- [Background] Pelletier JP, Martel-Pelletier J, Abramson SB. Osteoarthritis, an inflammatory disease: potential implication for the selection of new therapeutic targets. Arthritis Rheum. 2001 Jun;44(6):1237-47. doi: 10.1002/1529-0131(200106)44:63.0.CO;2-F. No abstract available. PMID 11407681
- [Background] Wang S, Wang H, Liu W, Wei B. Identification of Key Genes and Pathways Associated with Sex Differences in Osteoarthritis Based on Bioinformatics Analysis. Biomed Res Int. 2019 Dec 6;2019:3482751. doi: 10.1155/2019/3482751. eCollection 2019. PMID 31886203